CLINICAL TRIAL: NCT06048003
Title: Armenian National Registry of ST-elevation Myocardial Infarction,a Multicenter Prospective Observational Study With Biocollection
Brief Title: Armenian National Registry of Myocardial Infarction
Acronym: ARMI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Armenian Cardiologists Association (Other)
Collaborators: Santé Arménie French-Armenian Research Center (Other)
Responsible Party: Sponsor
Other Study IDs: ACA-2023001
Record Dates: First submitted 2023-09-15; First posted 2023-09-21 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-09

CONDITIONS: ST Elevation Myocardial Infarction
Keywords: STEMI; Myocardial infarction; acute coronary syndrome; CV mortality; biobanking
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Myocardial Infarction; Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No specific intervention — No specific intervention

SUMMARY:
This is a national, multicenter prospective observational study of patients presenting to hospitals in Armenia with STEMI diagnosis.

The main questions it aims to answer are:

* Determine the rate of in-hospital mortality for the patients with STEMI admitted to the participating hospitals.
* Compare short and long-term CV and all-cause mortality and hospitalization.
* Determine how professional guidelines are followed in real-world situations.

DETAILED DESCRIPTION:
Although the state program on primary percutaneous coronary intervention in ST elevated myocardial infarction, which was launched in 2015 helped to drastically decrease STEMI mortality rates, patients who had survived usually develop heart failure (HF) which leads to increased economic burden for the Armenian healthcare system.

The total duration of the study will be 24 months. The target number of the inclusion is 2500 patients. The follow-up period for enrolled patients will be 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patient (≥ 18 years of age),
2. Admitted to the participating centers for a STEMI within 48 hours of symptom onset: characterized by a rise and fall of cardiac markers (troponins) together with ST elevation in at least two contagious leads or LBBB.
3. Have given signed informed consent to participate in the study.

Non-Inclusion Criteria:

1. MI occurring ≤ 48 hours after PCI or CABG
2. The patient or the legal representative refused to sign the informed consent

Exclusion Criteria:

Withdrawal of the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The pre-screened population will consist of all patients >18 years old presenting acutely with suspected STEMI in the participating hospitals.
  Only patients with confirmed diagnosis of STEMI will be included in the registry, after informed consent signing.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Rate of the in-hospital mortality | During 5 to 7 days of hospitalization
  Determine the rate of the in-hospital mortality for the patients with STEMI admitted to the participating hospitals

SECONDARY OUTCOMES:
Cardiovascular mortality | 30 days and 12 months
  Compare short-term (30 days) and long-term (12 months) CV mortality depending on the management strategies.
All-cause mortality | 30 days and 12 months
  Compare short-term (30 days) and long-term (12 months) all-cause mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Hamlet G Hayrapetyan, Prof., Principal Investigator — Armenian Cardiologists Association
Locations (13):
- Armenia (13):
  - Vanadzor Medical Center, Vanadzor, Lori
  - Gyumri Medical Center, Gyumri, Shirak
  - French-Armenian Cardiovascular Center, Goris, Syunik
  - Heratsi Hospital Complex N1, Yerevan
  - Erebouni Medical Center, Yerevan
  - Aramyants Medical Center, Yerevan
  - Armenia Medical Center, Yerevan
  - Astghik Medical Center, Yerevan
  - Best Life Medical Center, Yerevan
  - Nork Marash Medical Center, Yerevan
  - Shengavit Medical Center, Yerevan
  - Surb Grigor Lusavorich Medical Center, Yerevan
  - Yerevan Scientific Medical Center, Yerevan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Armenian Cardiologists Association official website — https://armcardio.am/